CLINICAL TRIAL: NCT03394131
Title: Treatment of Carpal Tunnel in Rheumatoid Arthritis
Brief Title: ُEfficacy of Insulin Versus Hyalase Hydro-dissection of Median Nerve in Rheumatoid Arthritis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manal Hassanien, principle investigaror, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Hydrodissection of CT in RA
Record Dates: First submitted 2017-12-25; First posted 2018-01-09 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Treatment Resistant Carpal Tunnel in RA Patients
MeSH Terms: interventions — hylase; Hyaluronoglucosaminidase; Insulin; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hyalase (Experimental): injection and hydro-dissection of median nerve using hyaluronidase followed by 10 cc normal saline ultrasonic guided
  Interventions: Drug: Hylase
- Placebo (Placebo Comparator): injection and hydro-dissection of median nerve hydro-dissection using 10 cc saline injection ultrasonic guided
  Interventions: Other: saline
- Insilin (Active Comparator): injection and hydro-dissection of median nerve hydro-dissection using 10 IU insuline followed by 10 cc normal saline ultrasonic guided
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Hylase — hydro-dissection injection of median nerve inside carpal tunnel using hyalase and 10 cc saline
  Other Names: Hyaluronidase
  Arms: Hyalase
Drug: Insulin — hydro-dissection injection of median nerve inside carpal tunnel using 10 IU insulin and 10 cc saline
  Other Names: crystalline insulin
  Arms: Insilin
Other: saline — hydro-dissection injection of median nerve inside carpal tunnel using 10 cc saline
  Other Names: normal saline
  Arms: Placebo

SUMMARY:
Carpal tunnel syndrome (CTS) is a common peripheral entrapment neuropathy in Rheumatoid arthritis patients proved by nerve conduction studies and ultrasound parameters, this study aims to evaluate the effect of hydro-dissection using insulin versus hyalase versus saline, ultrasounic guided as an effective treatment

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is a common peripheral entrapment neuropathy in Rheumatoid arthritis patients proved by nerve conduction studies and ultrasound parameters, this study aims to evaluate the effect of hydro-dissection of median nerve inside CT twice injections with interval 2 weeks using insulin and 10 cc saline versus hyalase and 10 cc saline versus 10 cc saline, ultrasounic guided as an effective treatment of CT

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis in remission

Exclusion Criteria:

* active Rheumatoid arthritis

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
pain intensity | 6 months
  Visual analog scale 0-100

SECONDARY OUTCOMES:
nerve conduction | 6 months
  sensory velocity
ultrasound | 6 months
  cross sectional area

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hassanien, MD, Principal Investigator — Assiut University
Locations (1):
- Manal Hassanien, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Yes
after complete recruiting of patients
Supporting Information: Study Protocol
Time Frame: 1 year